CLINICAL TRIAL: NCT01562587
Title: Pharmacokinetics of Single Bolus Dose of NovoSeven® in Paediatric and Adult Patients With Haemophilia A or B in a Non-Bleeding State
Brief Title: Pharmacokinetics of Single Bolus Dose of NovoSeven® in Paediatric and Adult Patients With Haemophilia A or B in a Non- Bleeding State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F7HAEM-1503
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Haemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adults (Experimental)
  Interventions: Drug: activated recombinant human factor VII
- Paediatric (Experimental)
  Interventions: Drug: activated recombinant human factor VII

INTERVENTIONS:
Drug: activated recombinant human factor VII — A single bolus dose is administered. Injected intravenously
  Arms: Adults
Drug: activated recombinant human factor VII — A random order of a low/high dose of single dose is administered during two PK-assessment periods separated by a washout period of 48 hours to one month. Injected intravenously
  Arms: Paediatric

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to determine the pharmacokinetics of activated recombinant human factor VII (NovoSeven®) in haemophiliac patients in a non-bleeding state.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years and congenital haemophilia A or B male with severe FVIII or FX deficiency +/-inhibitors
* Age between 3-12 years and congenital haemophilia A or B male with record of inhibitors

Exclusion Criteria:

* Known hypersensitivity to activated recombinant human factor VII or any of its components
* Known clinical relevant coagulation diseases or insufficiencies other than congenital haemophilia
* Clinical manifestation of HIV (human immunodeficiency virus) and/or protease inhibitor treatment
* Clinical manifestation of active/recent bleeding
* Administration of coagulation factor preparations within 24 hours of NovoSeven trial product dose administration
* Body Mass Index (BMI) outside normal range
* Known abuse of elicit drugs and/or alcohol
* Renal insufficiency
* Hepatic disease
* Cardiovascular disease
* Any disease or condition which, judged by the Investigator, could imply a potential hazard to the patient, interfere with the trial participation or trial outcome

Ages: 3 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2002-09; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Area under the concentration curve from 0-12 hours

SECONDARY OUTCOMES:
CL, the total body clearance
Cmax, the maximum concentration
tmax, the time to maximum concentration
t1/2, the terminal half-life
Area under the concentration curve from time 0-infinity
Vss, the apparent volume of distribution at steady state
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (8):
- Germany (2):
  - Novo Nordisk Investigational Site, Bremen
  - Novo Nordisk Investigational Site, Frankfurt
- Novo Nordisk Investigational Site, Athens, Greece
- Italy (2):
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Milan
- Novo Nordisk Investigational Site, Madrid, Spain
- United Kingdom (2):
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Oxford

REFERENCES:
- [Result] Villar A, Aronis S, Morfini M, Santagostino E, Auerswald G, Thomsen HF, Erhardtsen E, Giangrande PL. Pharmacokinetics of activated recombinant coagulation factor VII (NovoSeven) in children vs. adults with haemophilia A. Haemophilia. 2004 Jul;10(4):352-9. doi: 10.1111/j.1365-2516.2004.00925.x. PMID 15230949
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com